CLINICAL TRIAL: NCT06413901
Title: TIP Repair of Distal Penile Hypospadias Using Rapidly Absorbable Braided Vs Slowly Absorbable Monofilament Sutures: A Prospective, Randomized Controlled Study
Brief Title: TIP Repair of Distal Penile Hypospadias Using Rapidly Absorbable Braided Vs Slowly Absorbable Monofilament Sutures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelghany, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-421-2023
Record Dates: First submitted 2024-05-05; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Hypospadias Repair

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vicryl group (Experimental): TIP hypospadias repair
  Interventions: Procedure: TIP
- PDS group (Experimental): TIP hypospadias repair
  Interventions: Procedure: TIP

INTERVENTIONS:
Procedure: TIP — TIP hypospadias repair

SUMMARY:
Objective:

To study the effect of tubularizing the urethral plate in DPH in children using 2 different absorbable suture materials, rapidly absorbable, braided 6/0 Vicryl and slowly absorbable monofilament 6/0 Polydioxanone, on complication rates.

Patients and methods:

A prospective, randomized controlled study conducted at the Urology Department, Cairo University Specialized Pediatric Hospital, Abou El Reesh, between September 2021 and September 2022. A total of 69 boys aged between 8 and 120 months with DPH were randomly divided into 2 groups: group(A) Vicryl included 39 boys and group(B) PDS included 30 boys. All boys were uncircumcised with no chordee and were primary repairs. TIP was the surgical technique used by a single pediatric urologist. Follow up was performed in outpatient clinic at 7 days, 1, 3, 6 and 12 months postoperatively. The complications and reoperation rates for both groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* Any child(aged from 6m to 12 years old) with distal penile hypospadias (DPH) ( uncircumcised, without chordae, with good penile size and urethral plate(candidates for T.I.P repair)

Exclusion Criteria:

* reccurent cases,
* circumcised cases
* other types of hypospadias rather than DPH,
* presence of chordae,
* poor urethral plate

Ages: 6 Months to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
complication rate | one year
  urethrocutaneous fistula, wound infection, wound dehiscence, overall complications, and reoperation rates

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt